CLINICAL TRIAL: NCT00749424
Title: CORONARY BIFURCATIONS: APPLICATION OF THE CRUSHING TECHNIQUE USING SIROLIMUS-ELUTING STENTS - The "CACTUS" Trial
Brief Title: The Study of the Crushing Technique Application Using SES in Coronary Bifurcations.
Acronym: CACTUS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cordis US Corp. (Industry)
Responsible Party: Hans-Peter Stoll, MD, Cordis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRDIT 00-01/03
Record Dates: First submitted 2008-09-08; First posted 2008-09-09 (Estimated); Last update posted 2010-02-04 (Estimated); Status verified 2010-02

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): crushing technique
  Interventions: Device: SES
- 2 (Active Comparator): provisional T stenting technique
  Interventions: Device: SES

INTERVENTIONS:
Device: SES — CYPHER SELECT™ Sirolimus-eluting Balloon-expandable Coronary Stent
  Arms: 1
Device: SES — CYPHER SELECT™ Sirolimus-eluting Balloon-expandable Coronary Stent
  Arms: 2

SUMMARY:
The objective of this study is to compare the safety and effectiveness of two different approaches to treat bifurcational lesions with CYPHER SELECT™ Sirolimus-eluting Balloon-expandable Coronary Stent , Cordis Corp): a) the "crushing" technique to stent both branches vs. b) a provisional T stenting technique of the side branch.

DETAILED DESCRIPTION:
This is a prospective, randomized study that will be conducted at up to 5 centers in Italy. All patients who meet the eligibility criteria will be treated with the Cypher SelectTM Stent and Stent Delivery System (SDS). Patients will have repeat angiography at six months, with clinical follow-up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Is a male or non-pregnant female patient >= 18 years of age [NOTE: Females of child-bearing potential must have a negative pregnancy test];
2. Has a diagnosis of angina pectoris as defined by Canadian Cardiovascular Society Classification (CCS I, II, III, IV) OR unstable angina pectoris (Braunwald Classification B&C, I-II) OR has documented silent ischemia;
3. Has at least TIMI I coronary flow in both the main and side branches;
4. Involves a single treatment of a de novo bifurcation lesion in native coronary arteries of patients with single or multivessel disease; patients with multiple lesions can be included only if other lesions treated during the index procedure are successfully treated prior to the treatment of the bifurcation lesion;
5. Has a true bifurcation lesion defined as stenosis > 50% in both the main branch and the ostium of the side branch;
6. Has a maximum treatable main or side branch lesion length <=28 mm;
7. Has a main branch vessel that is >= 2.5 mm and <= 3.5 mm in diameter by on-line QCA proximal to the bifurcation;
8. Has a side branch vessel that is >= 2.25 mm and <= 3.5 mm in diameter by on-line QCA;
9. Is an acceptable candidate for coronary artery bypass surgery (CABG);
10. Is willing to comply with the specified follow-up evaluation;
11. The patient or legally authorized representative must provide written informed consent prior to the procedure.

Exclusion Criteria:

1. Patient has experienced a Q-wave or non-Q-wave myocardial infarction with documented elevation of CK levels > 2 times normal or CK-MB levels > 3 times normal within the preceding 24 hours and/or the CK and CK-MB enzymes remain above normal at the time of treatment;
2. Has unstable angina classified as Braunwald A I-III, B&C III;
3. Has a bifurcation lesion in a non protected left main;
4. Has an ejection fraction <= 35%;
5. Has known allergies to the following: aspirin, clopidogrel bisulfate (Plavix) and ticlopidine (Ticlid), heparin, or sirolimus;
6. Has a known serious allergy to contrast media or stainless steel that cannot be managed medically;
7. Has impaired renal function (creatinine > 3.0 mg/dl);
8. There is presence of thrombus in the bifurcation lesion;
9. Has a target lesion with excessive tortuousity unsuitable for stent delivery and deployment;
10. Has a totally occluded vessel;
11. Is the recipient of a heart transplant;
12. Has a significant medical condition which in the investigator's opinion may interfere with the patient's optimal participation in the study;
13. Is currently participating in an investigational drug or another device study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2004-01; Primary Completion 2005-05 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Major Adverse and Cardiac Events (MACE) | 6 and 12 months post-procedure

SECONDARY OUTCOMES:
Minimal lumen diameter (MLD) | 6 months
Percent diameter stenosis (%DS) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Colombo, MD, PhD, Principal Investigator — Fondazione Centro San Raffaele del Monte Tabor
Locations (1):
- Fondazione Centro San Raffaele del Monte Tabor, Milan, Italy

REFERENCES:
- [Result] Colombo A, Bramucci E, Sacca S, Violini R, Lettieri C, Zanini R, Sheiban I, Paloscia L, Grube E, Schofer J, Bolognese L, Orlandi M, Niccoli G, Latib A, Airoldi F. Randomized study of the crush technique versus provisional side-branch stenting in true coronary bifurcations: the CACTUS (Coronary Bifurcations: Application of the Crushing Technique Using Sirolimus-Eluting Stents) Study. Circulation. 2009 Jan 6;119(1):71-8. doi: 10.1161/CIRCULATIONAHA.108.808402. Epub 2008 Dec 22. PMID 19103990